CLINICAL TRIAL: NCT00493662
Title: Cross-Over Evaluation of Two Lubricating Eye Drops
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 5310
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid; Sodium Chloride; sodium phosphate

INTERVENTIONS:
Drug: Polyethylene Glycol 400 0.4%
Drug: Propylene Glycol 0.3%
Drug: 0.15% sodium Hyaluronate
Drug: sodium chloride
Drug: sodium phosphate monobasic

SUMMARY:
To evaluate the efficacy of two lubricating eye drops for the treatment of dry eye signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 yrs or older
2. Males or females
3. Any race or ethnic background
4. Patients with present ocular surface discomfort and a SESoD score of at least 2

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Contact lens use on day of examination.
3. Corneal ectasia.
4. Current use of Restasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tom Kislan, OD, Principal Investigator — Hazleton Eye Specialists
Locations (1):
- Hazleton Eye Specialists, Hazleton, Pennsylvania, United States